CLINICAL TRIAL: NCT07208617
Title: Efficacy Superiority Trial of Red Light Myopia Control Device Based on LED Light Source
Brief Title: Development of Bioluminescent Myopia Prevention and Control Instrument and Evaluation of Its Effect on Myopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Ying Jie, Dr, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BeijingTH LED
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-09

CONDITIONS: Myopia
Keywords: Myopia; Red-light; LED light
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED red-light (Experimental)
  Interventions: Device: RED-light device using LED light source
- control (Sham Comparator): Fake light, with a light source power that is one-tenth of that of real LED light
  Interventions: Device: Control

INTERVENTIONS:
Device: RED-light device using LED light source — The light source type of red light is LED light source.
  Arms: LED red-light
Device: Control — Fake light, with a light source power that is one-tenth of that of real LED light
  Arms: control

SUMMARY:
Based on the Tongren Myopia and Amblyopia Therapeutic Apparatus (a 650nm low-level red-light device) developed by the research team in the previous phase, the device was modified by replacing the light source with LED light. Subsequently, a population study was conducted to evaluate its efficacy and safety in myopia prevention and control.

ELIGIBILITY:
Inclusion Criteria:

* Willing to use myopia treatment devices based on LED light sources or fake light sources Aged 6-18 years old For both eyes, the myopic spherical equivalent refraction after cycloplegic computerized refraction: -0.50D to -6.00D, and astigmatism ≤ 2.50D Spherical equivalent anisometropia of both eyes ≤ 2.50D Corrected visual acuity (for both near and far) ≥ 1.0 Intraocular pressure (IOP) 10-21mmHg No active ocular inflammation, no history of ocular trauma, no history of ocular surgery, and no ocular or systemic organic diseases that affect visual changes Voluntarily participate in this project and sign the informed consent form The subject has not used other myopia control methods in the past six months Have records of refractive error and axial length measurements six months before enrollment

Exclusion Criteria:

* Subjects with systemic diseases or immune diseases that affect compliance, such as tumors, heart diseases (including those with implanted electronic devices in the body, such as cardiac pacemakers), severe liver and kidney diseases, epilepsy, and autoimmune diseases Subjects with mental illnesses that affect the implementation of the intervention measures in this trial Subjects with refractive media opacity (corneal lesions, lens opacity, etc.) or ocular diseases: macular diseases, moderate to severe dry eye, corneal diseases, cataracts, vitreoretinal diseases, infectious conjunctivitis, uveitis, optic nerve damage, congenital optic nerve dysplasia, or other ocular diseases Subjects allergic to cycloplegics Other circumstances where the researcher deems it inappropriate for the subject to participate in the trial for safety reasons or in the interest of the patient

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 206 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Axial length | Baseline and 6-month follow-up
  Key parameter monitoring myopia progression
Spherical equivalent error | Baseline and 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No